CLINICAL TRIAL: NCT03972254
Title: Feasibility of Using Telepractice to Provide Modified Interaction Guidance as an Intervention Tool for Caregivers and Their Child With Autism
Brief Title: Feasibility of Using Telepractice to Provide Modified Interaction Guidance.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H2019:105
Record Dates: First submitted 2019-05-13; First posted 2019-06-03 (Actual); Last update posted 2022-01-12 (Actual); Status verified 2021-12

CONDITIONS: Autism Spectrum Disorder
Keywords: Modified Interaction Guidance
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Intervention Model Description: This study is a mixed methods feasibility study using a single-subject research design and qualitative description.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Caregivers and their child will interact for 10 minutes while being observed and videotaped. Psychoeducation will be provided and goal setting will occur to ensure dyad specific relationship gains are made.
  Interventions: Behavioral: Modified Interaction Guidance

INTERVENTIONS:
Behavioral: Modified Interaction Guidance — The main steps in the procedure are to have the family identify the primary concern they are facing, highlight the strengths that the family already has in place and expand on those strengths, convey/impart caregiving and societal norms, and offer other perspectives (McDonough, 2004). The goal of this therapy is to engage the family to take an active role in the construction of their overall treatment. The individualized treatment approach focuses and builds on existing strengths.

SUMMARY:
The purpose of this study is to determine the feasibility of using telepractice to provide Modified Interaction Guidance (MIG) to caregivers and their child with autism. MIG as an intervention to improve attachment for children with autism and their primary caregiver.

DETAILED DESCRIPTION:
The process objectives target focus on1) recruitment, 2) retention, 3) engagement with tools, 4) time demand on dyads, and 5) eligibility criteria.

The resource assessment objectives include: 1) equipment and internet accessibility 2) communication methods, and 3) timelines.

The management assessment objectives address: 1) ethical standards, 2) researcher qualifications and 3) data storage and collection.

Finally, when looking at the scientific assessment, the objectives relate to: 1) Is use of a concurrent multiple baseline single-subject design feasible with this population? 2)capturing dyad needs, 3) burden levels, and 4) safety protocols.

This study will evaluate the above listed dimensions of feasibility using a embedded mixed methods approach that incorporates both a single-subject design and qualitative data gathered throughout the research process and post intervention individual interviews.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of autism spectrum disorder
2. Child between the ages of 24-60 months
3. First born child
4. No physical or medical conditions that affect the child's ability to participate in the activities that are part of the intervention process
5. Ability to follow simple verbal directions in English
6. No current plan to initiate any treatment alternatives during the study period
7. Willingness to participate in a -week intervention with a frequency of once a week
8. Adults are primary caregiver
9. Under age of 35
10. Speak English
11. Minimum grade 5 schooling
12. Access to a computer and broadband wired or wireless (3G or 4G/LTE) internet connection?

Exclusion Criteria:

* Participants (both child and adult) will be excluded from the present study if they were deemed low functioning
* child is not the first-born child
* child already receiving ABA treatment
* parents have a history of mental illness

Ages: 10 Months to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 8 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Parenting Interactions with Children Checklist of Observations Linked to Outcomes (PICCOLO) | 4 weeks
  Serves as an observational tool to determine parental abilities in four specific domains; Affection, Responsiveness, Encouragement and Teaching.

SECONDARY OUTCOMES:
Goal Attainment Scale (GAS) | Immediately right before and after the Intervention
  Used to evaluate client specific goals. When goals are established by the client, the goals are then evaluated and measured by client specific criterion.

OTHER OUTCOMES:
Parent Sense of Competency (PSOC) | Baseline and 2 weeks post intervention.
  Measures parent's feelings of self-esteem and satisfaction of the ability in a parenting role. The PSOC is a 17 item scale, with 2 subscales. Each item is rated on a 6 point Likert scale anchored by 1 = "Strongly Disagree" and 6 = "Strongly Agree". A higher score indicates a higher parenting sense of competency.

CONTACTS AND LOCATIONS:
Overall Officials: Megan Land McCarthy, Bsc OT, Principal Investigator — University of Manitoba
Locations (1):
- College of Rehabilitation Sciences, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: No